CLINICAL TRIAL: NCT03988868
Title: The Effect of End-tidal Carbon Dioxide Level on the Optic Nerve Sheath Diameter Measured by a Transorbital Ultrasonography in Pediatric Patients
Brief Title: The Effect of End-tidal Carbon Dioxide Level on the Optic Nerve Sheath Diameter in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1904-053-1027
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia, General
Keywords: optic nerve sheath diameter; end-tidal carbon dioxide; trans-orbital ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Because the optic nerve is surrounded by the cerebrospinal fluid, increase / decrease in the intracranial pressure can be examined by an increase / decrease in the optic nerve sheath diameter (ONSD). Non-invasive trans-orbital ultrasonography has been used to measure the ONSD and shown to be useful in differentiating patients with increased intracranial pressure (> 20 cmH2O).

Arterial carbon dioxide partial pressure (PaCO2) is closely related to cerebral blood flow. According to the textbook, an increase in PaCO2 in the range of PaCO2 = 25 mmHg to PaCO2 = 75 mmHg can cause a change in intracranial pressure by proportionally increasing cerebral blood flow. Because end-tidal CO2 partial pressure (ETCO2) reflects PaCO2, a significant correlation may be expected between the ETCO2 and the ONSD.

Previous studies in adult patients showed that ONSD was sensitively increased / decreased according to short-term hypercapnia (ETCO2 = 50mmHg) or hypocapnia (ETCO2 = 30mmHg) for 10 minutes and normalized at normal ETCO2 (40mmHg). Therefore, the reactivity of the ONSD according to the change of the ETCO2 was confirmed in adult patients.

In normal pediatric patients, ONSD is expected to respond to changes in ETCO2. However, no previous study has confirmed this. In addition, the reactivity of ONSD was not studied in neonates and infants with open fontanelle.

In this study, the investigators will performed trans-orbital ultrasonography in pediatric patients with normal intracranial intracranial pressure aged 18 years or younger scheduled for surgery under general anesthesia. The ONSD will be measured at three ETCO2 levels; 35mmHg, 40mmHg, and 45mmHg.

DETAILED DESCRIPTION:
Induction of general anesthesia and endotracheal intubation will be performed with standard electrocardiography, non-invasive blood pressure, heart rate, pulse oximetry, and ETCO2 monitoring.

The ONSD will be measured at three different ETCO2 levels (35mmHg, 40mmHg, and 45mmHg). Each ETCO2 levels will be maintained within +-2mmHg for 3 minutes.

A high frequency linear probe will be used to get the images of optic nerve sheath and the diameter (ONSD) will be measured at 3 mm from the papillary segment in the transverse plane. Mean arterial pressure and heart rate will be recorded during ONSD measurements. The open or closure of Fontanelle will be examined after ONSD measurements.

The ONSD and OND measurements will be performed by two independent researchers who do not participate in ultrasound examination using stored images.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years of age who are under general anesthesia
* Mechanical ventilation by endotracheal intubation
* Supine position during surgery

Exclusion Criteria:

* Disease including eyeball or orbit
* Infection or trauma around the eyes
* Difficult to access the eyes during surgery (Ophthalmologic surgery, neurosurgery, otorhinolaryngology surgery, etc.)
* Patients with abnormal intracranial pressure abnormality (trauma, brain tumors, hydrocephalus, intracranial pressure control shunt, craniosynostosis..)
* Laparoscopic surgery, Thoracoscopic surgery
* Cerebrovascular disease such as Moyamoya disease
* Hypotension
* Atelectasis, pneumothorax, pleural effusion, pneumonia, wheezing or crackle before surgery
* History of adverse reaction to ultrasound gel or Tegaderm (3M Canada, London, Ont., Canada) for eyeball protection

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All ASA grade I-II pediatric patients with no evidence of increased intracranial pressure under 18 years of either gender undergoing surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | 1 weeks
  Optic nerve sheath diameter (ONSD) measured at three ETCO2 levels(35mmHg, 40mmHg, and 45mmHg) by transorbital ultrasonography

SECONDARY OUTCOMES:
Mean arterial pressure | 1 weeks
  Mean arterial pressure during ONSD measurements
Heart rate | 1 weeks
  Heart rate during ONSD measurements
Eyeball diameter | 1 weeks
  Eyeball diameter by transorbital ultrasonography
Open Fontanelle | 1 weeks
  Open of the Fontanelle by palpation
Age | 1 weeks
  Age
Sex | 1 weeks
  Sex
Weight | 1 weeks
  Weight
Height | 1 weeks
  Height
BMI | 1 weeks
  BMI

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD.PhD., Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le A, Hoehn ME, Smith ME, Spentzas T, Schlappy D, Pershad J. Bedside sonographic measurement of optic nerve sheath diameter as a predictor of increased intracranial pressure in children. Ann Emerg Med. 2009 Jun;53(6):785-91. doi: 10.1016/j.annemergmed.2008.11.025. Epub 2009 Jan 23. PMID 19167786
- [Background] Wang LJ, Chen LM, Chen Y, Bao LY, Zheng NN, Wang YZ, Xing YQ. Ultrasonography Assessments of Optic Nerve Sheath Diameter as a Noninvasive and Dynamic Method of Detecting Changes in Intracranial Pressure. JAMA Ophthalmol. 2018 Mar 1;136(3):250-256. doi: 10.1001/jamaophthalmol.2017.6560. PMID 29392301
- [Background] Dinsmore M, Han JS, Fisher JA, Chan VW, Venkatraghavan L. Effects of acute controlled changes in end-tidal carbon dioxide on the diameter of the optic nerve sheath: a transorbital ultrasonographic study in healthy volunteers. Anaesthesia. 2017 May;72(5):618-623. doi: 10.1111/anae.13784. Epub 2017 Feb 8. PMID 28177116